CLINICAL TRIAL: NCT05010837
Title: Effect of Kinesio Taping on Waist-to-hip Ratio, Abdominal Muscle Strength and Body Image Concerns in Postpartum Females.
Brief Title: Effect of KT Taping on Waist-to-hip Ratio, Abdominal Strength and Body Image Concerns in Postpartum Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TehreemJabir
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Postpartum Disorder
Keywords: waist circumference; waist to hip ratio; body image; post partum; exercise
MeSH Terms: conditions — Puerperal Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping with abdominal exercises (Experimental): Kinesio taping will be applied along with abdominal exercises.
  Interventions: Other: Kinesio taping with abdominal exercises
- Abdominal Exercises (Active Comparator): Only abdominal exercises will be administered to the participants.
  Interventions: Other: Abdominal exercises

INTERVENTIONS:
Other: Kinesio taping with abdominal exercises — Experimental group was given kinesio taping along with abdominal exercises. Kinesio taping was applied in I-band technique. the first band is applied on rectus abdominis from origin to insertion starting from pubic symphysis till the xiphoid process. the second band is applied bilaterally on the left and right side external oblique muscles.
  Abdominal exercises consist of 2-3 sets of 8 to 12 repetitions of head lift with bracing, head lift with pelvic tilt, pelvic clock, bridging, knee rolling and deep breathing exercises for 1 to 4 weeks.
  From 5 to 8 weeks Same abdominal exercises with 5 sets and 15 to 20 repetitions were performed along with kinesio taping.
  Arms: Kinesio taping with abdominal exercises
Other: Abdominal exercises — Abdominal exercises consist of 2-3 sets of 8 to 12 repetitions of head lift with bracing, head lift with pelvic tilt, pelvic clock, bridging, knee rolling and deep breathing exercises for 1 to 4 weeks.
  From 5 to 8 weeks Same abdominal exercises with 5 sets and 15 to 20 repetitions were performed.
  Arms: Abdominal Exercises

SUMMARY:
This study is aimed at determining the effect of kinesio taping on waist to hip ratio, abdominal muscle strength and body image concerns in postpartum females.

DETAILED DESCRIPTION:
Post Caesarian section there is abdominal weakness and an increase in fat ratio. There is a significant decrease in strength of abdominal muscles and an increase in fat ratio after the C section. Common increase in abdominal circumference in postpartum females and its long term outcomes like women health orders change in body shape and dissatisfaction is arising very commonly in society. Body Image Concern Inventory scale is used to assess dysmorphic concern of body. This study will work on the effects of Kinesiotaping which will be easily applicable and increase muscle activation along with abdominal exercises to regain lost muscle strength and tightening of loose skin. This tapping technique has a therapeutic effect on muscles and easily available in the rehabilitation department. Nowadays it is becoming very common, easily available, and regarded by physiotherapists as a method to support, rehabilitate and stimulate some physiological processes. This study aims at determining rehabilitative treatment to reduce waist circumference in post partum females.

ELIGIBILITY:
Inclusion Criteria:

* Prima parous females, eight weeks post-partum.
* Females with both vaginal delivery and C section.

Exclusion Criteria:

* Females who received previous abdominal or spinal surgeries.
* Females having infection in sutures.
* Females having abdominal hernia, skin sensitivity
* Females having moderate to severe Diastasis Recti (IRD more than 3 finger width).
* Neurological impairment affecting muscle performance.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Study is focused on postpartum females.
Enrollment: 24 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
waist to hip ratio | 8th week
  Changes from baseline waist circumference was measured using a non-elastic measuring tape was used perpendicular to the long axis of the body and horizontal to the floor at end of normal expiration at anatomic landmarks including midpoint between the lowest rib (below) and iliac crest (above). Hip Circumference was also measured around the largest parts of the hips. The waist-to-hip ratio was calculated by dividing the waist circumference by hip circumference. The scores were measured at baseline and after 8 weeks of intervention.

SECONDARY OUTCOMES:
Body Image concerns Inventory | 8th week
  changes from baseline Body image concerns were measured using body image concerns inventory. A brief questionnaire for assessment of dysmorphic concerns consisting of 19 points based on 5 points scale interpreting 1 never and 5 always. This scale indicates concerns relating to appearance, behavior, and social attitude. A highly useful, precise, and less time taking assessment regarding body concerns. Scores range from 19 to 95. where higher scores represent higher level of dysmorphic concerns.
Double leg lowering test | 8th week
  Changes from baseline double leg lowering test was used to assess abdominal strength. Participant lies supine with arms across chest, examiner raises patients lower leg vertically, procedure will be explained. Blood pressure cuff placed at pelvis level inflated at 40 mmHg. Participants instructed to lower both legs with the extended knee from the vertical position down while keeping the pelvis in the posterior tilting position, and the pressure cuff used as feedback to try to maintain the starting inflated pressure. During the test if the pressure on the cuff reduces the test is stopped and the angle is measured using goniometer from table. the strength is graded as poor for 75-90 degree from table, fair (3) for 46-75 degree from the table, Good (4) 16-45 degrees from the table and Normal (5/5) 0-15 degrees from the table

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Asia general hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohamed H, Yousef A, Kamel HE, Oweda K, Abdelsameaa G. Kinesio Taping and Strength Recovery of Postnatal Abdominal Muscles after Cesarean Section. Egyptian Journal of Physical Therapy 2020 Dec 15; 4(1):13-9.
- [Background] AcharryN, Kutty RK. Abdominal exercise with bracing, a therapeutic efficacy in reducing diastasis-recti among postpartum females Int J Physiother Res. 2015; (2):999-1005.
- [Background] Dave H, AratiMahishale MP. Effect of Structured Abdominal Exercise Programme on Diastasis of Rectus Abdominis Muscle in Postpartum Women-An Experimental Study (Doctoral dissertation, KLE University, Belagavi, Karnataka)
- [Background] Madly MM. Effect of Kinesio taping therapy on waist circumferences in postpartum women Journal of Medicine in Scientific Research. 2018 Jan 1; 1(1):4
- [Background] Gursen C, Inanoglu D, Kaya S, Akbayrak T, Baltaci G. Effects of exercise and Kinesio taping on abdominal recovery in women with cesarean section: a pilot randomized controlled trial. Arch Gynecol Obstet. 2016 Mar;293(3):557-65. doi: 10.1007/s00404-015-3862-3. Epub 2015 Sep 2. PMID 26329802
- [Background] Vispute SS, Smith JD, LeCheminant JD, Hurley KS. The effect of abdominal exercise on abdominal fat. J Strength Cond Res. 2011 Sep;25(9):2559-64. doi: 10.1519/JSC.0b013e3181fb4a46. PMID 21804427
- [Background] El-Mekawy HS, Eldeeb AM, El-Lythy MA, El-Begawy AF. Effect of abdominal exercises versus abdominal supporting belt on post-partum abdominal efficiency and rectus separation. InProceedings of World Academy of Science, Engineering and Technology 2013 Jan 1 (No. 73, p. 742). World Academy of Science, Engineering and Technology (WASET).
- [Background] Ghadakzadeh S, Ghazipour A, Khajeddin N, Karimian N, Borhani M. Body Image Concern Inventory (BICI) for identifying patients with BDD seeking rhinoplasty: using a Persian (Farsi) version. Aesthetic Plast Surg. 2011 Dec;35(6):989-94. doi: 10.1007/s00266-011-9718-8. Epub 2011 Apr 14. PMID 21491168
- [Background] Schulte-van Maaren YW, Giltay EJ, van Hemert AM, Zitman FG, de Waal MW, Van Rood YR, Carlier IV. Reference values for the Body Image Concern Inventory (BICI), the Whitely Index (WI), and the Checklist Individual Strength (CIS-20R): The Leiden Routine Outcome Monitoring Study. J Affect Disord. 2014 Aug;164:82-9. doi: 10.1016/j.jad.2014.03.013. Epub 2014 Mar 24. PMID 24856558
- [Background] Ptak A, Konieczny G, Stefanska M. The influence of short-term kinesiology taping on force-velocity parameters of the rectus abdominis muscle. J Back Musculoskelet Rehabil. 2013;26(3):291-7. doi: 10.3233/BMR-130382. PMID 23893144
- [Background] Littleton HL, Axsom D, Pury CL. Development of the body image concern inventory. Behav Res Ther. 2005 Feb;43(2):229-41. doi: 10.1016/j.brat.2003.12.006. PMID 15629752
- [Background] Benjamin DR, van de Water AT, Peiris CL. Effects of exercise on diastasis of the rectus abdominis muscle in the antenatal and postnatal periods: a systematic review. Physiotherapy. 2014 Mar;100(1):1-8. doi: 10.1016/j.physio.2013.08.005. Epub 2013 Oct 5. PMID 24268942
- [Background] Fu TC, Wong AM, Pei YC, Wu KP, Chou SW, Lin YC. Effect of Kinesio taping on muscle strength in athletes-a pilot study. J Sci Med Sport. 2008 Apr;11(2):198-201. doi: 10.1016/j.jsams.2007.02.011. Epub 2007 Jun 27. PMID 17588814
- [Background] El-Refaye GE, El Nahas EM, Ghareeb HO. Effect of kinesio taping therapy combined with breathing exercises on childbirth duration and labor pain: a randomized controlled trial. Bulletin of Faculty of Physical Therapy 2016 Jun; 21(1):23-31.
- [Background] Krause DA, Youdas JW, Hollman JH, Smith J. Abdominal muscle performance as measured by the double leg-lowering test. Arch Phys Med Rehabil. 2005 Jul;86(7):1345-8. doi: 10.1016/j.apmr.2004.12.020. PMID 16003662